CLINICAL TRIAL: NCT05530785
Title: An Exploratory Clinical Study of Radiotherapy Combined With Sintilimab Plus Bevacizumab Biosimilar in the Treatment of Unresectable Hepatocellular Carcinoma (uHCC) With Portal Vein Tumor Thrombus (PVTT)
Brief Title: Radiotherapy + Sintilimab + Bevacizumab Biosimilar for uHCC With PVTT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yongchang Zhang (Other)
Responsible Party: Sponsor-Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Organization: Hunan Province Tumor Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: uHCC with PVTT
Record Dates: First submitted 2022-08-27; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma Non-resectable
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): radiotherapy combined with sintilimab and bevacizumab biosimilar
  Interventions: Combination Product: radiotherapy combined with sintilimab and bevacizumab biosimilar

INTERVENTIONS:
Combination Product: radiotherapy combined with sintilimab and bevacizumab biosimilar — After signing informed consent, patients received sintilimab 200 mg intravenously on the first day of each cycle, Q3W; Bevacizumab biosimilar 7.5mg/kg was administered intravenously on the first day of each cycle, Q3W; Concurrent radiotherapy (single dose 3-8Gy, times 3-10, total dose 20-50Gy; The duration of radiotherapy was completed between the first administration of sintilimab and the second administration of bevacizumab, but it should be noted that the interval between before and after the administration of sintilimab and bevacizumab was at least 3 days.

SUMMARY:
This study was a prospective, single-arm, single-center, phase II exploratory clinical study. To investigate the efficacy and safety of radiotherapy combined with sintilimab and bevacizumab biosimilar in the treatment of unresectable hepatocellular carcinoma with portal vein tumor thrombus.

DETAILED DESCRIPTION:
After signing informed consent, patients received sintilimab 200 mg intravenously on the first day of each cycle, Q3W; Bevacizumab biosimilar 7.5mg/kg was administered intravenously on the first day of each cycle, Q3W; Concurrent radiotherapy (single dose 3-8Gy, times 3-10, total dose 20-50Gy; The duration of radiotherapy was completed between the first administration of sintilimab and the second administration of bevacizumab, but it should be noted that the interval between before and after the administration of sintilimab and bevacizumab was at least 3 days.

Patients will be performed enhanced CT/MRI every 2 months, to access the efficiency according to the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, undergoing enhanced CT/MRI. The overall survival (OS) was calculated as the time from enrollment until death or the last follow-up. Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 to access the safety.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatocellular carcinoma confirmed by histology/cytology, or patients with cirrhosis and meet the American Association for the Study of Liver Diseases (AASLD) clinical diagnostic criteria for HCC
2. Child-pugh grade A or B (≤7 points)
3. A score of 0-1 according to the Eastern Cooperative Oncology Group Physical Status Score (ECOG PS score);
4. Barcelona stage C; Inamicable for radical surgical resection or refusal of surgery without extra-hepatic metastases; Portal vein tumor thrombus (PVTT) was diagnosed by enhanced CT or enhanced MRI (type VP1 to VP3).
5. Had not received systemic therapy or radiotherapy before; Or disease progression after surgical resection or local treatment (without radiotherapy);
6. At least one measurable or evaluable lesion according to the response evaluation criteria for solid tumors, version 1.1 (RECIST V1.1); Or measurable lesions that had clearly progressed after local treatment (based on RECIST V1.1 criteria).
7. Patients with liver lesions and/or portal vein tumor thrombus lesions were treated with radiotherapy

Exclusion Criteria:

1. Previous histological/cytological diagnosis included fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, and other components.
2. The area to be treated had been previously treated with radiotherapy
3. Patients with extrahepatic metastases
4. Patients with tumor thrombus invasion into the superior mesenteric vein
5. Patients with inferior vena cava tumor thrombus.
6. Central nervous system metastases were present.
7. A history of hepatic encephalopathy, or a history of liver transplantation.
8. There are clinical symptoms of pleural effusion, ascites, or pericardial effusion that require drainage.
9. Patients with acute or chronic active hepatitis B or C with hepatitis B virus (HBV) DNA>2000IU/ml or 10^4 Copies/ml; Hepatitis C virus (HCV)RNA> 10^3 Copies/ml; Hepatitis B surface antigen (HbsAg) and anti-HCV antibody were both positive.
10. History of allergy to active ingredients and/or excipients of anti-PD-1 mab and anti-VEFG mab.
11. Other malignancies, except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix, were present within 5 years.
12. Bleeding events from esophageal or gastric fundus varices due to portal hypertension had occurred within the previous 6 months. Severe (G3) varicose veins were known to have been present on endoscopy within 3 months before the first dose. There was evidence of portal hypertension (including splenomegaly on imaging) and a high risk of bleeding as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response rate | up to 2 years from enrollment
  assessed according to the Response Evaluation Criteria in Solid Tumors RECIST Version 1.1, undergoing enhanced CT/MRI

SECONDARY OUTCOMES:
Objective Response rate, assessed according to the modified Response Evaluation Criteria | up to 2 years from enrollment
  assessed according to the modified Response Evaluation Criteria in Solid Tumors Version 1.1, undergoing enhanced CT/MRI
overall survival | up to 2 years from enrollment
  the time from enrollment until death or the last follow-up
number of participants with treatment-related adverse events | up to 2 years from enrollment
  number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Jia Luo, Professor, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No